CLINICAL TRIAL: NCT03044262
Title: Evaluation of the Influence of Output on Skin Covered by Newly Developed Adhesives
Brief Title: Evaluation of the Influence of New Adhesives of Output on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_07
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 7 (Experimental): This is a sub-study testing the effect of real output applied under two adhesive strips (standard adhesive strip and new adhesive strip) on the skin after 8 hours.
  Interventions: Other: Standard adhesive strip; Other: New adhesive strip

INTERVENTIONS:
Other: Standard adhesive strip — This is a standard adhesive strip (hydrocolloid) that is part of an ostomy device
Other: New adhesive strip — This is a newly developed adhesive strip that in the future might be part of an ostomy device

SUMMARY:
The study investigates the impact real output has on peristomal skin covered by a newly developed adhesive and a standard adhesive

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Have had an ileostomy for more than one year
4. Have intact skin on the area used in the evaluation
5. Has an ileostomy with a diameter up to (≤) 35 mm
6. Have a peristomal area accessible for application of patches/adhesive strips (assessed by investigating scientist)

Exclusion Criteria:

1. Currently receiving or have within the past 2 month received radio- and/or chemotherapy
2. Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
3. Are pregnant or breastfeeding
4. Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
5. Participating in other interventional clinical investigations or have previously participated in this evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
Trans epidermal water loss | 8 hours
  The condition of the skin (trans epidemeral water loss) is measured after removing the adhesive.

CONTACTS AND LOCATIONS:
Overall Officials: Lene Feldskov, M. Sci, Principal Investigator — R&D scientist
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No